CLINICAL TRIAL: NCT05600153
Title: Axillary Versus Primary Breast Approach for Second-stage Operation in Expander-Implant Breast Reconstruction
Brief Title: Axillary Versus Primary Breast Approach for Second-stage Breast Reconstruction
Acronym: AvBSR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Affiliated Hangzhou First People's Hospital, Zhejiang University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2022- 1451
Record Dates: First submitted 2022-10-12; First posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Breast Neoplasm Female; Breast Reconstruction; Wound Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- primary breast approach (Placebo Comparator)
  Interventions: Procedure: implant exchange operation
- axillary approach (Experimental)
  Interventions: Procedure: implant exchange operation

INTERVENTIONS:
Procedure: implant exchange operation — To perform implant exchange via axillary incision.

SUMMARY:
The goal of this clinical trial is to compare the safety of axillary or primary breast approach for second-stage operation in expander-implant breast reconstruction for breast cancer patients. The main question it aims to answer are: 1. if the wound related events, including wound dehiscence, infection, delayed healing is significant less often in patients receiving second stage operation via axillary approach compared with primary breast approach; 2. if the aesthetic outcome is comparable between patients receiving different approach for second stage operation. To answer these questions, the breast cancer patients have received nipple-sparing or skin-sparing mastectomy and had breast tissue expander insertion via breast incision, will be prospectively recruited, and randomized into two groups while receiving implant exchange operation: (1) operate via axillary incision; (2) operate via primary breast incision.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 + (inclusive)
* Female
* Invasive breast cancer or ductal carcinoma in situ was confirmed by preoperative pathology
* SSM/NSM (skin sparing/nipple and areola sparing mastectomy) combined with expander implantation has been performed within a year
* An incision on the surface of the breast is used to place an expander in the first-stage surgery
* There is no clinical or radiological evidence of distant metastasis
* Expander removal combined with prosthesis implantation is planned
* Able and willing to sign an informed consent

Exclusion Criteria:

* The first SSM/NSM combined expander implantation was performed via axillary approach
* Patients participate in other clinical trial, which could potentially affect their participation in this trial
* Adjuvant radiotherapy was planned post-operation
* Patient who is pregnant and lactating
* The expander is not sufficiently expanded pre-surgery (does not reach more than 90% of its volume)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of Wound healing within 7 days post-operation | up to 7 days post-operation
  Without one of the following conditions：wound dehiscence requiring local wound care or operative intervention, wound infection requiring antibiotics 24hours post-operation, or debridement, within 7 days of post-operation.

SECONDARY OUTCOMES:
other surgical complications | one year
  Including hematoma, seroma, nipple and areola Necrosis, implant exposure, implant removal, and cyst contracture, measured by Clavien-Dindo stage.
Breast Q score | one year
  The satisfaction of breast reconstruction of participants will be measured by Breast Q questionnaire 12 months post-operation. Breast-Q questionnaire is based on 6 dimensions: Physical health, mental health, sexual health, satisfaction with breast, satisfaction with surgical outcome, and satisfaction with medical care. The scores of each dimension are expressed as independent scores between 0 and 100 calculated by the Q Score system.
Length of incision | up to 7 days post-operation
  length of incision measured within one-week post-operation.
Pathological evaluation | through study completion
  A piece of scar tissue will be collected during surgery and embedded with paraffin, and pathological evaluation, including Masson staining, immune histochemistry of desmin, SMA, Ki67，TGFβ，Smad2/3，CTGF/CCN2，IL-6, IL-8，MMP-1，MMP-2，MMP-3，MMP-13，COL I，COLIII, COL-5. And the staining intensity will be measured by two independent pathologists.

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Anyone needs individual participant data should contact the main investigator via e-mail.